CLINICAL TRIAL: NCT01915277
Title: A Phase I Study of Dexmedetomidine Bolus and Infusion in Corrective Infant Cardiac Surgery: Safety and Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHN-DEX
Record Dates: First submitted 2013-07-30; First posted 2013-08-02 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Transposition of the Great Arteries; Tetralogy of Fallot; Ventricular Septal Defect
Keywords: Pediatric corrective cardiac surgery
MeSH Terms: conditions — Transposition of Great Vessels; Tetralogy of Fallot; Heart Septal Defects, Ventricular | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Neonate dosing cohort 1 (Experimental): Neonate dexmedetomidine dosing cohort 1
  Interventions: Drug: Dexmedetomidine
- Neonate dosing cohort 2 (Experimental): Neonate dexmedetomidine dosing cohort 2
  Interventions: Drug: Dexmedetomidine
- Neonate dosing cohort 3 (Experimental): Neonate dexmedetomidine dosing cohort 3
  Interventions: Drug: Dexmedetomidine
- Neonate dosing cohort 4 (Experimental): Neonate dexmedetomidine dosing cohort 4
  Interventions: Drug: Dexmedetomidine
- Neonate dosing cohort 5 (Experimental): Neonate dexmedetomidine dosing cohort 5
  Interventions: Drug: Dexmedetomidine
- Infant dosing cohort 1 (Experimental): Infant dexmedetomidine dosing cohort 1
  Interventions: Drug: Dexmedetomidine
- Infant dosing cohort 2 (Experimental): Infant dexmedetomidine dosing cohort 2
  Interventions: Drug: Dexmedetomidine
- Infant dosing cohort 3 (Experimental): Infant dexmedetomidine dosing cohort 3
  Interventions: Drug: Dexmedetomidine
- Infant dosing cohort 4 (Experimental): Infant dexmedetomidine dosing cohort 4
  Interventions: Drug: Dexmedetomidine
- Infant dosing cohort 5 (Experimental): Infant dexmedetomidine dosing cohort 5
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: Precedex, dexmedetomidine HCl

SUMMARY:
The purpose of this Phase I study is to determine the safety of a drug called dexmedetomidine (DEX) as part of a balanced general anesthetic and sedative strategy for neonates and infants undergoing corrective cardiac surgery that requires the use of cardiopulmonary bypass for congenital cardiac problems. This study will also design and validate a dosing schema for the use of DEX as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 0 to 180 days at the time of surgery.
2. Diagnosis of: D-transposition of the great arteries (with or without ventricular septal defect), or tetralogy of Fallot, or ventricular septal defect (with or without associated atrial septal defect and/or patent ductus arteriosus)
3. Scheduled for complete corrective two-ventricle surgical repair with cardiopulmonary bypass.

Exclusion Criteria:

* 1. Less than 37 completed weeks' gestational age at birth for the Neonatal age group (0-21 days); less than 36 completed weeks' gestational age at birth for the Infant age group (22-180 days).

  2. Enrollment in the PHN Collaborative Learning Study, if tetralogy of Fallot 91-180 days of age only.

  3. Known or suspected hepatic dysfunction; AST and ALT >3X upper limit of normal at the time of screening within 72 hours of operation.

  4. Known or suspected renal dysfunction; serum creatinine > 0.8 mg/dL after 7 days of age, >1.2 mg/dL if <7 days of age, within 72 hours of operation.

  5. Preoperative administration of DEX or clonidine within 72 hours of operation.

  6. Major congenital anomaly(ies) outside the cardiovascular system that in the investigator's opinion would potentially affect safety or pharmacokinetics.

  7. Preoperative central nervous system injury resulting in clinical signs and symptoms: coma, seizures, hemiparesis.

  8. Planned period of deep hypothermic circulatory arrest. 9. History of second or third degree heart block. 10. Sinus or junctional bradycardia below 80 BPM sustained for greater than 15 minutes within 72 hours of operation. 11. Junctional rhythm sustained for greater than 15 minutes within 72 hours of operation.

  12. Hypotension defined as mean arterial blood pressure below 35 mm Hg for 0-21 day old neonatal patients, and below 40 mm Hg for 22-180 day old infant patients sustained for greater than 15 minutes within 72 hours of operation.

  13. History of cardiac arrest or ECMO cannulation.

Max Age: 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
The occurrence of a safety event that is possibly, probably or definitely related to DEX administration | Within 4 hours after DEX adminstration
  The occurrence of any of the following that is possibly, probably, or definitely related to DEX administration:
  * Bradycardia
  * Heart block
  * Junctional rhythm
  * Hypotension
  * Excessive sedation
  * Cardiac arrest or ECMO cannulation
  * Serious Adverse Event (SAE)
  Both the DEX dose, and DEX exposure will be assessed for associations with the primary outcome.

SECONDARY OUTCOMES:
Plasma concentration of DEX | Intraoperatively and up to 36 hours post-operatively
  Plasma concentrations of dex obtained intraoperatively and up to 36 hours post-operatively will be used to create drug dosing models. These models will then be evaluated to determine how effective they are at achieving targeted plasma concentration levels.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Zuppa AF, Nicolson SC, Wilder NS, Ibla JC, Gottlieb EA, Burns KM, Stylianou M, Trachtenberg F, Ni H, Skeen TH, Andropoulos DB; Pediatric Heart Network Investigators. Results of a phase 1 multicentre investigation of dexmedetomidine bolus and infusion in corrective infant cardiac surgery. Br J Anaesth. 2019 Dec;123(6):839-852. doi: 10.1016/j.bja.2019.06.026. Epub 2019 Oct 14. PMID 31623840